CLINICAL TRIAL: NCT02256254
Title: SIMOX - A Randomized, Double-blinded, Placebo Controlled Study of Simvastatins Possible Effect on Oxidative Stress on Healthy Volunteers
Brief Title: SIMOX - Induction of Oxidative Stress
Acronym: SIMOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Klinisk Biokemisk Afdeling (Unknown); Klinisk farmakologisk Afdeling (Unknown); Sektion for Biomedicin Institut for Veterinær Patobiologi (Unknown)
Responsible Party: Principal Investigator, Henrik Enghusen Poulsen, Professor MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2014-647
Record Dates: First submitted 2014-09-22; First posted 2014-10-03 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Oxidative Stress
Keywords: Oxidative stress; Simvastatin
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): 2 Simvastatin capsules of 20 mg every evening for 14 days
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): 2 placebo capsules every evening for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 2 Simvastatin capsules of 20 mg every evening for 14 days
  Arms: Simvastatin
Drug: Placebo — 2 placebo capsules every evening for 14 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate if use of simvastatin is associated with the level of oxidative stress in humans. The association is examined by comparing changes in oxidative stress in a group treated with simvastatin with the change in a placebo group. The study is a randomized-based, double-blinded placebo-controlled study. Each treatment group consists of 20 healthy male volunteers who consume simvastatin or placebo over 14 days. The induction of oxidative stress is measured by 8-oxoguanosine and 8- oxodeoxyguanosine, isolated from urine. A t-test will be performed to compare drug treatment with placebo. The results will be published.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* healthy men
* 18-50 years
* BMI: 18-30

Exclusion Criteria:

* Total cholesterol less than 3 mmol/L
* Use of natural and herbal medicines that is affected/affects simvastatin:

anion exchangers, amiodarone, amlodipine, ciclosporin, clarithromycin, colchicine, danazol, diltiazem, erythromycin, fibrates, fluconazole, fusidin acid, grape fruit juice, HIV protease inhibitors, itraconazole, ketoconazole, nefazodone, niacin, posaconazole, rifampicin, telithromycin, verapamil, vitamin K-antagonists, voriconazole

* following diseases: a Coronary vascular disease b Renal insufficiency c Hepatic insufficiency d heart failure e Previous heart arrythmia f Hypokalaemia g Low blood pressure h hyperthyroidism i muscular toxicity j galactose intolerants k Lapp Lactase deficiency l Glucose/galactose-malabsorption m Psychiatric disorder
* allergies towards any of the tested medicine
* intake of narcotics within 2 months prior to trial
* intake of supplements within 2 months prior to trial

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of 8-oxoguanosine (nmol/24h) | Change from Baseline after fourteen days of treatment
Urinary excretion of 8-oxodeoxyguanosine (nmol/24h) | Change from Baseline after fourteen days of treatment

SECONDARY OUTCOMES:
Malondialdehyde | Change from Baseline after fourteen days of treatment
Vitamin C | Change from Baseline after fourteen days of treatment
Vitamin E | Change from Baseline after fourteen days of treatment
Biopterin | Change from Baseline after fourteen days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Enghusen Poulsen, Professor MD, Principal Investigator — Department head
Locations (1):
- Department of Clinical Pharmacology, Copenhagen, Denmark